CLINICAL TRIAL: NCT06560801
Title: Randomized Clinical Study to Analyse the Effects of Dapagliflozin on Renal Morphology and Renal Perfusion in Patients With Impaired Renal Function One Year After Kidney Transplantation
Brief Title: Dapagliflozin on Renal Morphology and Renal Perfusion in Patients One Year After Kidney Transplantation
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Roland E. Schmieder, Prof. Dr. med., University of Erlangen-Nürnberg Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dapa-TxV1.0
Record Dates: First submitted 2024-08-12; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Drug: dapagliflozin, other: standard of care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin (Active Comparator): Dapagliflozin + standard of care
  Interventions: Drug: Dapagliflozin 10mg Tab
- Standard of care (No Intervention): standard of care only

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — Randomization will take place at visit 1 to either the group receiving standard care and dapagliflozin or standard care only.
  Arms: Dapagliflozin

SUMMARY:
The aim of this study is to observe the mechanisms of dapagliflozin on the renal interstitial tissue and renal perfusion. For this purpose, renal transplanted patients as an excellent model of CKD and high cardiovascular risk (similar to patients in DAPA-CKD study) are included in this study.

The objectives of the study are to analyze the effects of dapagliflozin on renal morphology and renal perfusion in patients with impaired renal function one year after kidney transplantation. This is a randomized (1:1), single centre clinical study. Each patient will be randomly assigned in an unblinded fashion to 10 mg Dapagliflozin or not 9 months after transplantation. At least 48 patients will be randomized and included. The routine renal biopsy taken one year after kidney transplantation will allow us to determine the morphological integrity of peritubular fibroblasts, interstitial inflammatory cell density and investigate markers of inflammation, oxidative stress and nitic oxide synthase expression (iNOS).

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) has a high prevalence globally and is a global health concern. CKD is associated with increased risks of cardiovascular morbidity, mortality and decreased quality of life in all stages of the disease. Most patients with CKD die of cardiovascular events in earlier stages before end-stage renal disease develops.

For the last years, renin-angiotensin-aldosterone blockade agents (ACEi/ARBs) were the only treatment available for managing CKD in both native and kidney transplant patients. Recently, sodium-glucose transport protein 2 inhibitors (SGLT2i) emerged as a new class of therapeutics for diabetic CKD, non-diabetic proteinuric CKD, and heart failure with and without type 2 diabetes mellitus (T2DM) in patients with native kidneys.

Dapagliflozin (SGLT2i) has been shown to be cardio- and nephroprotective in patients with and without T2DM. The DAPA-CKD trial found that patients with CKD treated with dapagliflozin had a lower risk of the primary composite outcome of a sustained decline in the estimated glomerular filtration rate (eGFR) of at least 50%, end-stage kidney disease, or death from renal or cardiovascular causes than patients who were assigned to receive placebo. Similar results have been confirmed by other SGLT2i in 2022 (Empagliflozin; EMPA-KIDNEY trial). In April 2021, Dapagliflozin became the first SGLT2i to be approved by the Food and Drug Administration (FDA) for the treatment of chronic kidney disease (CKD) regardless of diabetic status.

The anti-hyperglycaemic and anti-hypertensive effects of Dapagliflozin have been extensively studied and demonstrated in a number of clinical trials as well as in a real-world care setting. Previously,the investigators have demonstrated treatment with dapagliflozin in patients with T2DM improved diabetic control and reduced blood pressure (BP) in comparison to placebo. Furthermore, the drug was capable of reducing hyperperfusion of retinal capillaries and minimizing arteriole remodelling, factors that contribute to the progression of diabetic retinopathy, known to be linked with diabetic nephropathy. However, the precise mechanisms of its nephroprotective potential are still under discussion and needs to be elucidated.

Recently, the investigators described the intrarenal and glomerular hemodynamics of SGLT2i assessed by the clearance technique. SGLT2-inhibition impacts predominantly on post glomerular site, decreases renal vascular resistance and preserves renal perfusion in patients with type 2 diabetes and, thereby preserve renal function.

Vascular, glomerular and tubular effects of SGLT2i are discussed based on experimental and rarely on human data. Since the SGLT2 transporter has a high oxygen demand, relative hypoxia occurs in the renal interstitial tissue, with morphological changes of the fibroblasts (impairing erythropoietin production). In addition, the high glucose milieu in the interstitium also causes increased oxidative stress and triggers inflammatory responses that may cause increased glomerular permeability (despite upregulation of nitric oxide synthesis) and interstitial fibrosis. The aim of this study is to observe the mechanisms of dapagliflozin on the renal interstitial tissue (histology, urinary and serum markers indicative of histological integrity) and renal perfusion. For this purpose, renal transplanted patients as an excellent model of CKD and high cardiovascular risk (similar to patients in DAPA-CKD study) are included in this study. In addition, the investigators obtain clinical data of SGLT2i administered in patients after kidney transplantation.

Up to date the use SGLT2i appear to be safe in patients after renal transplantation based on data from pilot studies. However, renal transplanted patients were not included in the large preapproval randomized placebo-controlled trials. So, treatment with SGLT2i in renal transplanted patients with CKD is not obligatory. Recently, a review has been published summarizing the potential benefits and concerns of these agents in the context of kidney transplantation. In summary, the frequency of reported adverse effects in kidney transplant recipients does not appear to exceed those found in non-transplant patients or in kidney transplant recipients in the absence of SGLT2i therapy. In particular, the incidence of urinary tract infections with SGLT2i were consistent with previously reported incidence rates of the same and there were no reported incidences of Fourier's gangrene.

Along with the histological parameters, the investigators assess parameters of the renal circulation including total renal perfusion, separate cortical and medullary renal perfusion and renal vascular resistance in this cohort using arterial spin labeling magnetic resonance imaging (ASL-MRI). Of note, we have demonstrated that renal perfusion assessed by ASL-MRI is valid, plausible and reliable.

Several prospective studies reported a closer relation of organ damage with central (aortic) as opposed to peripheral (brachial) systolic blood pressure (BP), and central systolic BP was found to be independently associated with cardiovascular morbidity and mortality. In accordance, central pulse pressure has been repeatedly found to independently predict cardiovascular morbidity and mortality in various study cohorts. Further-more, prospective data have now been published showing that the forward and backward (reflected) wave amplitude predict independently cardiovascular complications. New advanced technology allows us to assess different vascular parameters. Previously, the investigators could demonstrate that the SGLT2i empagliflozin and dapagliflozin improved parameters of vascular function and arterial stiffness and decreased central (aortic) pulse and systolic pressures (i.e. afterload of the left ventricle) in patients with T2DM. Our results provided evidence for the concept that the better cardiovascular and renal outcomes observed with dapagliflozin and empagliflozin in the outcome studies are related to improved vascular function. In this study, these parameters are assessed to find out if the above mentioned results can be confirmed in patients after renal transplantation.

Our hypothesis is that dapagliflozin exerts beneficial effects on renal morphology, intrarenal inflammation and oxidative stress in patients with CKD. Moreover, improve vascular parameters and renal perfusion. Our approach would add valuable information for our pathophysiological understanding of the nephroprotective mechanisms of dapagliflozin in patients with CKD. In addition, the investigators obtain clinical data with respect to safety and effectiveness of SGLT2i administered in patients after kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients aged between 18 and 75 years
* Patients with renal transplant having a stable eGFR, who are in stable condition, 9 months after transplantation, irrespective of their diabetes status
* Females of child bearing potential must be using adequate contraceptive precautions
* Females of childbearing potential or within two years of the menopause must have a negative urine pregnancy test at screening visit
* Informed consent (§ 40 Abs. 1 Satz 3 Punkt 3 AMG) has to be given in written form

Exclusion Criteria:

* Type 1 diabetes mellitus.
* HbA1c > 10%
* Use of SGLT-2 inhibitor within the past 2 months
* Any history of stroke, transient ischemic attack, instable angina pectoris, or myocardial infarction within the last 3 months prior to study inclusion.
* eGFR <25 ml/min/1.73m² (CKD-EPI Formula).
* Uncontrolled arterial hypertension (RR > 180/110 mmHg).
* Congestive heart failure (CHF) NYHA stage IV.
* Recurrent urinary tract infections (bacterial or fungal)
* Severe disorders of the gastrointestinal tract or other diseases which interfere the pharmacodynamics and pharmacokinetics of the drug.
* Significant laboratory abnormalities such as SGOT or SGPT levels more than 5 x above the upper limit of normal range.
* Antihypertensives are allowed but should be kept stable throughout the study period.
* Statins and other antihyperlipidemic drugs are allowed but should be kept stable throughout the study period.
* Drug or alcohol abusus
* Pregnant or breast-feeding patients
* Patients with contraindications to MRI

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
renal morphology - fibroblasts | 3 months after randomization
  integrity of peritubular fibroblasts (PDGFRα) assessed from the routine one year follow up biopsy of the renal transplant
renal morphology - inflammation | 3 months after randomization
  markers of inflammation (example CD3, CD68, CD163) in the interstitium from the routine one year follow up biopsy of the renal transplant
renal morphology - oxidative stress | 3 months after randomization
  markers of oxidative stress (Nox1, 8-OHdG) in the interstitium assessed from the routine one year follow up biopsy of the renal transplant

SECONDARY OUTCOMES:
mRNA Expression profile of transcripts | 3 months after randomization
  mRNA Expression profile of transcripts relevant in renal transplantation using the Human Organ Transplant Panel of NanoString including 770 genes.
renal perfusion | 3 months after randomization
  renal perfusion of the renal transplant measured by ASL-MRI
central (aortic) systolic pressurepulse pressure | 3 months after randomization
  central (aortic) systolic pressure and pulse pressure
pulse pressure | 3 months after randomization
  pulse pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center (CRC), Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No